CLINICAL TRIAL: NCT03464799
Title: Does Immunotherapy Have a Role in the Management of Endometriosis?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Hale GOKSEVER CELIK, Principal investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: KanuniSSRTH
Record Dates: First submitted 2018-01-09; First posted 2018-03-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: immunohistochemical staining — immunohistochemical staining

SUMMARY:
Pathological specimens of 40 women that had been operated for endometriosis will be included in this study. These tissues will be stained with a marker named as PDL-1 in pathological examination. "programmed cell death (PD-1)" is expressed on T cells. The immunotherapies in which antibodies against these PD-1 and its ligands (PDL-1) have been used are accepted as very effective in the treatment of many cancers. If these ligands can be shown in the endometriosis, it will be an important step for the treatment of endometriosis.

DETAILED DESCRIPTION:
40 women who had been operated for endometriosis between 2013 and 2014 will be included in this study. Pathological specimens will be stained with an immunohistochemical marker named as PDL-1. "programmed cell death (PD-1)" is a protein containing 288 aminoacids and expressed on T cells. It was shown on apoptotic cells in earlier times, but then it has been understood that its physiologic role is not cell death. The upregulation of PD-1 is a result of the activation of T cells and it is necessary for the termination of immune response. PD-L1 is a ligand for PD-1. The immunotherapies in which antibodies against these PD-1 and its ligands (especially PDL-1) provides significant improvements in many cancers such as melanoma. Evidence about the role of these ligands in endometriosis will be an important step in its management.

ELIGIBILITY:
Inclusion Criteria:

* patients operated for endometriosis between 2013 and 2014
* pathological examinations proving the diagnosis of endometriosis

Exclusion Criteria:

* patients operated for cysts other than endometriosis

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients operated for endometriosis
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
immunohistochemical staining | 6 months
  immunohistochemical staining with PD-L1